CLINICAL TRIAL: NCT04954664
Title: Lateral Ridge Augmentation Using Allograft Bone Particles Hydrated With or Without Recombinant Human Platelet-Derived Growth Factor: A Clinical and Histological Randomized Controlled Trial
Brief Title: Ridge Augmentation Using Allograft Particles Hydrated With or Without Recombinant Human Platelet-Derived Growth Factor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hussein Basma, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300007719; UAB Periodontology (Other: UAB)
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Dental Implant; Bone Loss
Keywords: New bone; Dental implants
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The calibrated, trained, masked-examiner (who is unaware of which Group the patient is randomized), will be masked and available during the entire duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft particles hydrated with rhPDGF (Experimental): Allograft particles should be hydrated with GEM21S for 20 minutes prior to grafting. The graft sites will be covered with a resorbable barrier membrane.
  Interventions: Biological: Allograft particles hydrated with rhPDGF
- Allograft particles hydrated in a conventional way with saline. (Active Comparator): Allograft particles should be hydrated with saline for 20 minutes prior to grafting. The graft sites will be covered with a resorbable barrier membrane.
  Interventions: Biological: Allograft particles hydrated in a conventional way with saline.

INTERVENTIONS:
Biological: Allograft particles hydrated with rhPDGF — Allograft particles should be hydrated with GEM21S for 20 minutes prior to grafting. The graft sites will be covered with a resorbable barrier membrane.
  Arms: Allograft particles hydrated with rhPDGF
Biological: Allograft particles hydrated in a conventional way with saline. — Allograft particles should be hydrated with saline for 20 minutes prior to grafting. The graft sites will be covered with a resorbable barrier membrane
  Arms: Allograft particles hydrated in a conventional way with saline.

SUMMARY:
This study will compare two techniques to achieve increase in ridge dimensions as a preparation for dental implants using a resorbable barrier membrane and bone particulate allogenic graft hydrated with saline or a growth factor called Recombinant Human Platelet-Derived Growth Factor (rhPDGF).

DETAILED DESCRIPTION:
This is a prospective, randomized, and examiner-only-masked study. It is designed to clinically compare the use of bone particulate allograft hydrated with rhPDGF vs bone particulate allograft hydrated with saline, for patients who were planned to receive dental implants but presented with deficient bone ridges. This investigation of two techniques to achieve increase in ridge dimensions as a preparation for dental implants using a resorbable barrier membrane and bone particulate allogenic graft hydrated with saline or a growth factor called Recombinant Human Platelet-Derived Growth Factor (rhPDGF).

In two arms, bone core biopsies will be harvested at time of implant placement 4 months following ridge augmentation grafting. These 2x8mm bone cores will then undergo histological and histomorphometrical analyses to determine qualitative and quantitative healing differences between in both study arms.

Clinical measurements are gathered at 2 time points (grating and implant placement) at all defects and will be compared for differences.

Cone beam computed tomography (CBCT) initial scans are conducted immediately following prior to ridge augmentation and second scans obtained prior to implant placement both arms. These types of Cone Beam CT scans as well as conventional dental x-rays are valuable treatment planning tools that are commonly used in modern-day implant dentistry. The scans and the x-ray images are also used to monitor the health of tissues surrounding implants and to make sure that the implant remains securely implanted into the jawbone over time.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Need for implants to replace missing tooth or teeth in at least one quadrant of the mouth.
* Insufficient alveolar ridge width for endosseous implant placement defined as 5mm or less as determined by bone sounding and cone beam computed tomography (CBCT) scan.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Patient is a poor compliance risk (i.e., poor oral hygiene, history of alcohol or drug abuse)
* Vertical loss of bone at edentulous ridge.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative histomorphometric evaluation of new bone formation 4 months after GBR | From baseline to 4 months
  To quantify the distribution of the different tissues (new bone, soft tissue, residual graft and artifact) after 4 months of healing. Hence, the primary outcome will be the new bone formation, defined as the percentage of new bone area in the histomorphometric sections.

SECONDARY OUTCOMES:
Quantitative two- and three-dimensional radiographic comparison of dimensional changes 4 months using cone beam computed tomography (CBCT) and a virtual implant planning software, coDiagnostiX™ | From baseline to 4 months
  quantification of bone width gain after ridge augmentation. both clinically using a caliper to measure the ridge width before and after ridge augmentation and also radiographically using a software that superimpose before and after CBCT to calculate the difference which basically leads to amount of bone gain.

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No